CLINICAL TRIAL: NCT03600558
Title: Efficacy of Fludarabine, Cytarabine and G-CSF (FLAG Regimen) for the Treatment of Patients With Acute Myeloid Leukemia (AML)
Brief Title: Efficacy of FLAG Regimen for the Treatment of Patients With AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, ZhongHong Shao, head of department of Hematology, Tianjin Medical University General Hospital
Other Study IDs: Handong
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute
Keywords: FLAG
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The long-term efficacy of chemotherapy in patients with acute myeloid leukemia (AML) has been significantly improved in recent years. The combination of anthracycline plus cytarabine (Ara-C) has been a standard induction regimen for patients with AML. However, the optimal consolidation therapy after induction chemotherapy has not reached a consensus. The FLAG regimen consisting of fludarabine and high-dose cytarabine combined with G-CSF which is one of the first-line consolidation treatment options for relapsed and refractory AML. This study conducted a retrospective analysis of the intensive treatment of AML with the FLAG regimen from January 2007 to May 2018 in our hospital to evaluate the efficacy of the FLAG regimen. To provide the basis for the choice and timing of treatment for patients with AML treated with the FLAG regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 year old
* De novo or secondary leukemia.
* Treated with FLAG regimen

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort, using medical charts of AML patients treated with the FLAG regimen from January 2007 to May 2018
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  For evaluating the FLAG effect, OS was defined from consolidation randomization to death from any cause (censored at last contact).

SECONDARY OUTCOMES:
Relapse-free survival | 2 years
  Relapse Free Survival defined as the time from onset of FLAG treatment for AML to the first event (death or relapse).
Severe adverse events | 45 days
  Severe adverse events during consolidation treatment
Complete Remission Rate | 2 months
Event-Free Survival Rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China